CLINICAL TRIAL: NCT00513708
Title: Helping Alcoholics Link to Substance Abuse Treatment Programs After Being in the Hospital for Detoxification
Brief Title: Facilitating Aftercare for Alcohol Detox Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Richard Blondell, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLO-NIAAA-015616; K23AA015616 (NIH)
Record Dates: First submitted 2007-08-07; First posted 2007-08-09 (Estimated); Results first posted 2011-03-08 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Alcohol Abuse; Alcohol Dependence
Keywords: Detoxification; Treatment
MeSH Terms: conditions — Alcoholism | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment As Usual (TAU) (No Intervention): Treatment as Usual (TAU): Participants randomized to this arm will receive "usual care" (i.e., pharmacotherapy to manage alcohol withdrawal, counseling and referral to treatment or self-help) during medically managed inpatient detoxification.
- Motivational Enhancement Therapy (MET) (Experimental): Participants randomized to this arm will receive "usual care" (i.e., pharmacotherapy to manage alcohol withdrawal, counseling and referral to treatment or self-help) during inpatient detoxification plus a 60-minute Motivational Enhancement Therapy (MET) session delivered by a trained professional.
  Interventions: Behavioral: Motivation Enhancement Therapy (MET)
- Peer-delivered Twelve Step Facilitation (Experimental): Participants randomized to this arm will receive "usual care" (i.e., pharmacotherapy to manage alcohol withdrawal, counseling and referral to treatment or self-help) during inpatient detoxification plus a 60-minute Peer-delivered Twelve Step Facilitation (P-TSF)session delivered by individuals from a common self-help program.
  Interventions: Behavioral: Peer-Twelve Step Facilitation (P-TSF)

INTERVENTIONS:
Behavioral: Motivation Enhancement Therapy (MET) — Participants assigned to this arm will receive a 60-minute MET intervention in addition to "usual care" while hospitalized for detoxification.
  Other Names: Brief Intervention
  Arms: Motivational Enhancement Therapy (MET)
Behavioral: Peer-Twelve Step Facilitation (P-TSF) — In addition to "usual care" while hospitalized for detoxification, participants assigned to this arm will receive a 60-minute visit by peers who are "recovering from alcoholism" and who are active in 12-step oriented self-help programs.
  Other Names: "12th Step Calls"
  Arms: Peer-delivered Twelve Step Facilitation

SUMMARY:
The purpose of this study is to determine whether peer visits (known as "12th Step Calls") and professional counselors (using "Motivational Enhancement Therapy") are effective helping alcoholics link to substance abuse treatment programs after being in the hospital for detox.

DETAILED DESCRIPTION:
For those with an alcohol use disorder, the decision to seek detoxification treatment often represents a desire or willingness to change drinking behavior. This gives clinicians with the opportunity to intervene and improve the lives of these individuals. Even patients admitted involuntarily or who have been coerced may be amenable to change. Therefore, inpatient alcohol detoxification treatment offers an opportunity to prepare these patients for and link them with aftercare treatment.

Unfortunately, clinicians have little to guide them on how the current standard of care for alcohol detoxification might be improved. Improvement in clinical practice is ideally driven by clinical research, but there is little recent published information to guide the development of evidence-based pharmacological or psychological practices or interventions in detoxification settings. As a result, alcohol detoxification treatment has changed little over the past 25 years.

Taken as a whole, the literature suggests that the outcomes of inpatient detoxification are less than optimal. A limited number of published studies suggest that a majority of these patients are not linked to any aftercare following inpatient detoxification treatment and return to drinking within a few weeks of hospital discharge. However, there is some evidence to suggest that interventions, performed while the patient is hospitalized, could encourage patients to initiate involvement in aftercare (i.e., professional treatment and/or mutual self-help following hospitalization) and to decrease drinking or initiate abstinence. Motivational Enhancement Therapy and Twelve-Step Facilitation are two interventions that show promise.

The study proposed in this study addresses this issue by testing two brief interventions, Motivation Enhancement Therapy (MET) and Peer-Twelve Step Facilitation (P-TSF, also known as "12th Step Calls"), which have shown potential to enhance initiation of a period of abstinence and engagement in treatment and/or self-help programs among alcohol detoxification patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female inpatients 18 years of age or older.
* Participants will have a current DSM-IV diagnosis of alcohol abuse or dependence.
* Able to understand/speak English
* Participants will have signed a witnessed informed consent.

Exclusion Criteria:

* Cognitive impairment (e.g., mental retardation)
* Participants who meet current DSM-IV criteria for bipolar disorder, schizophrenia, or dementia
* Participants who are homeless, without contact person
* Participants enrolled in a methadone maintenance treatment program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D. Blondell, MD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- Erie County Medical Center, Buffalo, New York, United States

REFERENCES:
- [Derived] Blondell RD, Frydrych LM, Jaanimagi U, Ashrafioun L, Homish GG, Foschio EM, Bashaw HL. A randomized trial of two behavioral interventions to improve outcomes following inpatient detoxification for alcohol dependence. J Addict Dis. 2011 Apr;30(2):136-48. doi: 10.1080/10550887.2011.554777. PMID 21491295

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment as Usual: Treatment as Usual (TAU): Participants randomized to this arm will receive "usual care" (i.e., pharmacotherapy to manage alcohol withdrawal, counseling and referral to treatment or self-help) during medically managed inpatient detoxification.
- Motivational Enhancement Therapy: Participants randomized to this arm will receive "usual care" (i.e., pharmacotherapy to manage alcohol withdrawal, counseling and referral to treatment or self-help) during inpatient detoxification plus a 60-minute Motivational Enhancement Therapy (MET) session delivered by a trained professional.
Period: Overall Study
Arm/Group | Treatment as Usual | Motivational Enhancement Therapy | Peer-delivered Twelve Step Facilitation
Started | 50 | 50 | 50
Completed | 46 | 46 | 46
Not Completed | 4 | 4 | 4
Not completed — Lost to Follow-up | 4 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual | Motivational Enhancement Therapy | Peer-delivered Twelve Step Facilitation | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 48 | 49 | 146
  >=65 years | 1 | 2 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.58 (9.92) | 44.96 (10.75) | 44.48 (12.36) | 45.34 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 25 | 33 | 78
  Male | 30 | 25 | 17 | 72
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: Linkage to Alcohol Behavioral Therapy Counseling (i.e., "Aftercare")
Description: Linkage to alcohol behavioral therapy counseling (i.e., "aftercare") was defined as: arriving for the first outpatient chemical dependency counseling visit, being admitted to an inpatient or residential chemical dependency treatment facility, or attending at least one meeting of a help-help program such as Alcoholics Anonymous.
Time Frame: 1 month
Population: There were 50 participants in each arm. Per protocol, the "number of participants analyzed" represents the number that had outcome data (i.e, "linked to aftercare" or "not linked to aftercare") available at the 30-day follow-up.
Measure: Number; unit: participants
Arm/Group | Treatment as Usual | Motivational Enhancement Therapy | Peer-delivered Twelve Step Facilitation
Number analyzed (Participants) | 44 | 44 | 43
participants | 36 | 36 | 32

2. Secondary Outcome: Relapse to Drinking
Description: Relapse to drinking was defined as the consumption of one or more standard drinks (approximately 12 grams of ethanol)during the first 30 days following discharge from the inpatient detoxification unit. The date of discharge was considered to be "Day 1."
Time Frame: 30 days
Population: There were 50 participants in each arm. Per protocol, the "number of participants analyzed" represents the number that had outcome data (i.e, "relapse" or "no relapse") available at the 30-day follow-up.
Measure: Number; unit: participants
Arm/Group | Treatment as Usual | Motivational Enhancement Therapy | Peer-delivered Twelve Step Facilitation
Number analyzed (Participants) | 42 | 43 | 41
participants | 23 | 25 | 20

3. Secondary Outcome: Completed Inpatient Treatment
Description: Completion of inpatient treatment was defined as being admitted to and successfully discharged from an inpatient alcohol treatment program (e.g., a "28-day program"). Participants who left the inpatient program "against medical advice" or who received an "administrative discharge" were not considered to have successfully completed the inpatient program.
Time Frame: 90 days
Population: There were 50 participants in each arm; the "number of participants analyzed" represents the number of those 50 in each arm who were admitted to an inpatient treatment program (e.g., a "28-day program").
Measure: Number; unit: Participants
Arm/Group | Treatment as Usual | Motivational Enhancement Therapy | Peer-delivered Twelve Step Facilitation
Number analyzed (Participants) | 19 | 25 | 12
Participants | 15 | 21 | 9

ADVERSE EVENTS:
Time Frame: During the initial 30-day follow-up one participant expressed suicidal ideation, which was reported to the IRB. Participant recruitment was suspended for approximately 2 weeks until a new protocol was developed.
Description: The participant, who expressed suicidal ideation, was referred to a counseling program, which resolved the problem. The participant was stable at the 90-day follow-up. It was determined that the participant used suicidal ideation in an attempt to ask the research for a date to have coffee.
Arm/Group | Treatment as Usual | Motivational Enhancement Therapy | Peer-delivered Twelve Step Facilitation
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes